CLINICAL TRIAL: NCT07185984
Title: Functional Development and Clinical Validation of a Diagnostic Tool Based on Artificial Intelligence for the Assessment of Sperm Quality and the Selection of the Optimal In Vitro Fertilisation (IVF) Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Other Study IDs: 2407-VLC-156-MM
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Infertility (IVF Patients); Male Fertility; Sperm Selection
Keywords: Male infertility; Microfluidics; Artificial intelligence; Sperm quality
MeSH Terms: conditions — Infertility; Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRELIMINARY SPERM ANALISYS: Small aliquots of 100 fresh human semen samples will be analysed using the SwimCount™ Harvester system. The sperm variables analyzed will include concentration, motility (total and progressive), morphology, movement speed, and trajectory.
  Interventions: Diagnostic Test: Sperm sellection
- DIAGNOSIS TOOL VALIDATION: 100 additional fresh semen samples processed with the integrated microfluidics system (SwimCount™ Harvester) and the CASA system with artificial intelligence
  Interventions: Diagnostic Test: DIAGNOSIS TOOL

INTERVENTIONS:
Diagnostic Test: Sperm sellection — Small aliquots of 100 fresh human semen samples will be analysed using the SwimCount™ Harvester system, a CE-marked microfluidic technology patented by MCount and designed for routine clinical use.
  Groups: PRELIMINARY SPERM ANALISYS
Diagnostic Test: DIAGNOSIS TOOL — The diagnostic tool developed will be validated by analyzing small aliquots of 100 additional fresh semen samples processed with the integrated microfluidic system (SwimCount™ Harvester) and the CASA system with artificial intelligence. To evaluate the diagnostic efficiency of the tool, the results obtained from the semen quality analysis will be compared with those obtained from the analysis of these samples when processed using the reference technique, based on conventional methods employed by fertility specialists. Finally, to determine the effectiveness of the developed tool, the clinical results obtained from assisted reproduction treatment will be compared with the diagnosis predicted by the tool, with the aim of evaluating its predictive capacity.
  Translated with DeepL.com (free version)
  Groups: DIAGNOSIS TOOL VALIDATION

SUMMARY:
Infertility is a growing global health problem affecting millions of couples worldwide, with male infertility accounting for approximately half of all cases. In the physiological environment, sperm go through an exhaustive selection process in the female reproductive tract before reaching the oocyte. During this journey, progressive mobility and morphology are key parameters for achieving fertilisation. Therefore, before starting an assisted reproduction treatment, it is essential to analyse and process the semen sample to assess the fertile potential, select the most optimal sperm and determine the most appropriate treatment.

Conventional methods of semen processing, such as density gradient centrifugation (DGC) and Swim-up washing of motile sperm, have significant limitations. These include interobserver and interlaboratory subjectivity, as well as damage to sperm DNA caused by centrifugation. Alternatively, microfluidics, which simulates natural selection, allows higher counts of morphologically normal, progressive motile sperm to be obtained. On the other hand, the CASA (computer-assisted sperm analysis) system has improved the standardisation and quality of semen analysis. Furthermore, the incorporation of Artificial Intelligence (AI) into semen quality analysis represents a promising opportunity, as it improves efficiency, accuracy and standardisation, and has the potential to increase success rates in assisted reproduction treatments.

This project aims to develop an innovative AI-based diagnostic tool to address male infertility. The tool will integrate microfluidic technology and the CASA system to analyse semen quality, calculate fertilisation potential and recommend personalised treatments with an estimate of success. Trained with large volumes of biological and clinical data, it will provide a comprehensive and patient-specific diagnosis by identifying complex relationships between multiple variables. Finally, a comparative study will be conducted to evaluate laboratory indicators and clinical outcomes of cycles using this tool versus those using conventional methods.

ELIGIBILITY:
* Inclusion criteria:

  * Men between the ages of 18 and 50 who come to the clinic to undergo an ICSI cycle.
  * Men between the ages of 18 and 50 who come to the clinic to undergo an artificial insemination cycle.
  * All embryos will be placed in a time-lapse incubator.
  * All women over 18 years of age who have obtained a MII number greater than or equal to 2 in oocyte retrieval, without excluding couples from the oocyte donation programme.
  * All men and women with a previously known normal karyotype.
  * Informed consent (IC) provided and signed by patients.
* Exclusion criteria:

  * All women diagnosed with recurrent pregnancy loss.
  * All semen samples obtained by testicular biopsy.
  * All donor semen samples.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will include patients who attend the IVIRMA Valencia clinic for a cycle of artificial insemination or a cycle of ICSI and undergo sperm selection using the Harvester microfluidic technique.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Development of a Male Infertility Diagnosis Tool | 2 YEARS
  Tool development

SECONDARY OUTCOMES:
Prediction Capability Identification | 2 Years
  Measure of correlation between clinical data and tool prediction
Development of an AI algorithm | 2 years
  Development of an AI algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Meseguer, PhD, Principal Investigator — IVIRMA Valencia
Locations (1):
- IVI Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://linkinghub.elsevier.com/retrieve/pii/S0093691X13003555
- See also: Related Info — https://www.dovepress.com/some-of-the-factors-involved-in-male-infertility-a-prospective-review-peer-reviewed-article-IJGM
- See also: Related Info — https://linkinghub.elsevier.com/retrieve/pii/S0015028220307779
- See also: Related Info — https://linkinghub.elsevier.com/retrieve/pii/S0015028298001460